CLINICAL TRIAL: NCT00582803
Title: Adherence to Intensive Surveillance for Hereditary Breast Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Mark Robson, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 03-059
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: breast cancer; germline mutation; BRCA1; BRCA2; family history; genetic testing; unaffected women over age 25 who are at elevated risk for; breast cancer by virtue by a hereditary predisposition
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Women with strong family histories of breast cancer are at increased risk to have breast cancer. Women whose close relatives have had breast cancer often have more breast cancer screening than other women their age. To increase the chance that any breast cancer will be caught early, women at risk often take part in special screening programs. These programs involve more frequent visits to the doctor for breast exams, yearly mammography, and new types of exam like breast Magnetic Resonance Imaging (MRI). Studies are going on to find out whether these programs are better than standard screening. The purpose of this study is to find out how these programs impact women's quality of life. The study will also try to learn what factors make it hard to take part in the programs. We hope to be able to design new programs that are easier to follow.

DETAILED DESCRIPTION:
Women at risk for hereditary breast cancer are recommended to undergo intensive surveillance to maximize the likelihood of detecting the disease at an early, more curable, stage (Burke et al. 1997, Eisenger et al. 1998, Moller et al. 1999). Although the particular recommendations of different groups have varied, all suggest programs that incorporate clinical and radiographic screening performed more frequently than in the general population, beginning at a considerably younger age. Recent studies demonstrating the sensitivity of breast MRI have led several groups to incorporate this technology as an incremental (not replacement) modality, further increasing the intensity of the surveillance regimen. While data are beginning to accumulate regarding the effectiveness of aggressive surveillance, little is known about the ability and willingness of women to adhere to these rigorous schedules, nor about the psychosocial and economic costs of the programs. Based upon the Cognitive-Social Health Information Processing (C-SHIP)model (Miller, Shoda, Hurley 1996), we hypothesize that the ability to adhere to a proposed screening regimen will result from a complex and dynamic interaction between the nature of that regimen, events that can be expected to occur in the course of screening (such as abnormal results and practical barriers) and key psychological factors such as the individual's attentional style, affective state, perceived risk of cancer, cancer-specific worries, and beliefs regarding the effectiveness of screening. To test the hypothesis, we propose to prospectively study women with a hereditary risk for breast cancer participating in a structured surveillance program of monthly breast self-examination, semi-annual clinical examination and annual mammography, augmented by annual interval breast MRI.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 25 years or greater
* Genetic predisposition as defined by one of the following:

  * Known BRCA1 or BRCA2 mutation (deleterious or uncertain significance) OR
  * Untested first-degree relative of an individual with a known deleterious BRCA mutation OR
  * Unaffected first-degree relative of an affected individual within a hereditary breast-ovarian kindred in which no testing has been performed or testing is negative, defined as: 3 or more women in 2 generations affected with breast or ovarian cancer. Women with bilateral breast cancer and woman with both breast and ovarian cancer count as single individual AND 1 woman must be first-degree relative of the other two, or related to the other two through a male AND At least 1 woman affected with breast cancer before age 50 or ovarian cancer at any age
* Able to understand and complete English-language questionnaires
* Intend to receive clinical and radiographic follow-up at MSKCC

  * Women will not be excluded if they have previously received clinical and radiographic follow-up at either MSKCC or another institution.

Exclusion Criteria:

* Prior history of breast or ovarian cancer
* Contraindication to breast MRI examination (e.g. aneurysm clips, pacemaker, cochlear implant, severe claustrophobia, weight over 300 pounds) or to paramagnetic contrast (prior IgE-type allergic reaction, sickle cell anemia, renal failure)
* Pregnant or planning to begin attempts at conception within 1 year of enrollment. A negative serum β-hCG will not be required for study entry, nor for radiographic examination, as this test is not routinely performed before clinically indicated radiographic study.
* Unable for physical, psychological, or financial reasons to receive clinical and radiographic follow-up at MSKCC
* Concurrent medical or psychological conditions that, in the opinion of the attending physician or Principal Investigator, would place the subject at risk were she to participate

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: unaffected women over age 25 who are at elevated risk for breast cancer by virtue by a hereditary predisposition
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2003-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
cognitive-affective mediating units that are likely to be involved in health information processing and the execution of health-protective behavior | 5 years 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark Robson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org